CLINICAL TRIAL: NCT04008134
Title: CHoBI7 Trial: A Hospital Based Water, Sanitation and Hygiene Intervention for Households of Diarrheal Patients in Bangladesh
Brief Title: Cholera-Hospital-Based-Intervention-for-7-days
Acronym: CHoBI7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00006785; PR-15133 (Other: icddr,b)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cholera; Diarrhea; Stunting
Keywords: handwashing with soap; water treatment; behavior change; water, sanitation and hygiene
MeSH Terms: conditions — Cholera; Diarrhea; Growth Disorders

STUDY DESIGN:
Masking Description: Masking was not possible because the intervention included visible components including a handwashing station and a covered drinking water storage vessel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard recommendation (ORS) (No Intervention): Participants received the standard recommendation on oral rehydration solution use
- mHealth with no home visits (Experimental): Participants received the health facility delivery of CHoBI7, plus bi-weekly mHealth (voice and text) reminders for 12 months
  Interventions: Behavioral: CHoBI7 health facility program; Behavioral: CHoBI7 mHealth program
- mHealth with home visits (Experimental): Participants received the health facility delivery of CHoBI7, plus two home visits and bi-weekly mHealth (voice and text) reminders for 12 months
  Interventions: Behavioral: CHoBI7 health facility program; Behavioral: CHoBI7 mHealth program; Behavioral: CHoBI7 home visit program

INTERVENTIONS:
Behavioral: CHoBI7 health facility program — The CHoBI7 health facility program focuses on promoting handwashing with soap and water treatment to diarrhea patients and their household members during the one-week period after the patient is admitted to the health facility, when their household is at highest risk for diarrheal diseases. The CHoBI7 program includes: (1) a WASH pictorial module delivered by a health worker bedside to diarrhea patient and their household members in a health facility on handwashing with soap, water treatment, and safe water storage; and (2) a diarrhea prevention package containing chlorine tablets for water treatment, a soapy water bottle (water and detergent powder), a handwashing station, and a water vessel with a lid and tap for safe drinking water storage. Households are instructed to boil their water once their supply of chlorine tablets is completed.
  Arms: mHealth with home visits; mHealth with no home visits
Behavioral: CHoBI7 mHealth program — The CHoBI7 mHealth (mobile health) program targets five key behaviors: (1) preparing soapy water using water and detergent powder; (2) handwashing with soap at food and stool related events; (3) treating household drinking water using chlorine tablets during the one week high risk period after the diarrhea patient in the household was admitted to the health facility; (4) safe drinking water storage in a water vessel with a lid and tap; and (5) heating of household drinking water until it reaches a rolling boil after the one week high risk period. Participant households receive bi-weekly voice and text messages from the CHoBI7 mHealth program over a 12-month period. These mobile messages are sent using the VIAMO platform (www.viamo.io).
  Arms: mHealth with home visits; mHealth with no home visits
Behavioral: CHoBI7 home visit program — The CHoBI7 home visit program involves two, 30-minute home visits conducted during the week after the index diarrhea patient was recruited at the health facility. A health worker reinforces the content of the CHoBI7 health facility program in the participant's home.
  Arms: mHealth with home visits

SUMMARY:
The Cholera Hospital Based Intervention for 7 Days (CHoBI7) randomized controlled trial for transition to scale aimed to: (1) Develop and evaluate scalable approaches to integrate the CHoBI7 intervention into the services provided for hospitalized diarrhea patients at health facilities in Bangladesh; and (2) Evaluate the ability of the CHoBI7 intervention to lead to a sustained uptake of the promoted hand washing with soap and water treatment behaviors and significant reductions in diarrheal disease over time.

DETAILED DESCRIPTION:
The findings from the recent randomized controlled trial of The Cholera Hospital Based Intervention for 7 Days (CHoBI7) demonstrated that this intervention was effective in significantly reducing symptomatic cholera infections in intervention households, and had significant sustained impacts on hand washing with soap behaviors and improved water quality 12 months post intervention. Next steps to transition to scale were: (1) Develop and evaluate scalable approaches to integrate the CHoBI7 intervention into the services provided for hospitalized diarrhea patients at health facilities in Bangladesh; and (2) Evaluate the ability of the CHoBI7 intervention to lead to a sustained uptake of the promoted hand washing with soap and water treatment behaviors and significant reductions in diarrheal disease over time.

ELIGIBILITY:
Inclusion Criteria:

Diarrhea patients will be defined as patients having acute watery diarrhea three or more loose stools over a 24-hour period in the past three days. Diarrhea patients admitted to ICDDRB Dhaka Hospital or Mugda General Hospital will be eligible for the trial if:

1. have had 3 or more loose stools over the past 24 hours
2. plan to reside in Dhaka for the next 12 months
3. have no basin for running water in their home
4. have a child under five years of age in their household (including themselves) that produced a stool sample at baseline
5. have a working mobile phone in the household.

Household members of the diarrhea patient will be eligible for the trial if:

1. they have shared the same cooking pot and resided in the same home with the diarrhea patient for the last three days
2. plan to reside in their current household with the diarrhea patient for the next 12 months

Exclusion Criteria:

(1) Children in foster care will be excluded from all research study activities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2626 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Diarrhea prevalence among children under 2 years of age | 12 months
  Diarrhea prevalence among children under 2 years of age assessed by caregiver self report over a 12-month period
Diarrhea prevalence among children under 5 years of age | 12 months
  Diarrhea prevalence among children under 5 years of age assessed by caregiver self report over a 12-month period
Diarrhea prevalence among all household members | 12 months
  Diarrhea prevalence among all household members assessed by self report over a 12-month period

SECONDARY OUTCOMES:
Diarrhea prevalence among participants ages 5-9 years | 12 months
  Diarrhea prevalence among all household members ages 5-9 years assessed by self report over a 12-month period
Diarrhea prevalence among participants ages 10-18 years | 12 months
  Diarrhea prevalence among all household members ages 10-18 years assessed by self report over a 12-month period
Diarrhea prevalence among participants ages greater than 18 years | 12 months
  Diarrhea prevalence among all household members ages greater than 18 years assessed by self report over a 12-month period
Handwashing with soap | 12 months
  Household members handwashing with soap at food and stool related events assessed by 5-hour structured observation over a 12-month period
Household drinking water treatment | 12 months
  Households with stored drinking water samples without detectable E.coli (<1 colony forming units / 100 ml) assessed by unannounced household visits for sample collection of household stored drinking water over a 12-month period
Height-for-age among children under 2 years of age | 12 months
  Height, weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Height-for-age among children under 5 years of age | 12 months
  Height, weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate height-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age among children under 2 years of age | 12 months
  Height, weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-age among children under 5 years of age | 12 months
  Height, weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-age z-scores according to the World Health Organization child growth standards
Weight-for-height among children under 2 years of age | 12 months
  Height, weight and age measurements among children under 2 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards
Weight-for-height among children under 5 years of age | 12 months
  Height, weight and age measurements among children under 5 years of age assessed over a 12-month period were used to calculate weight-for-height z-scores according to the World Health Organization child growth standards

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] George CM, Monira S, Zohura F, Thomas ED, Hasan MT, Parvin T, Hasan K, Rashid MU, Papri N, Islam A, Rahman Z, Rafique R, Islam Bhuyian MS, Saxton R, Labrique A, Alland K, Barman I, Jubyda FT, Afroze F, Sultana M, Johura FT, Khan MAH, Tahmina S, Munmun F, Sack DA, Perin J, Alam M. Effects of a Water, Sanitation, and Hygiene Mobile Health Program on Diarrhea and Child Growth in Bangladesh: A Cluster-randomized Controlled Trial of the Cholera Hospital-based Intervention for 7 Days (CHoBI7) Mobile Health Program. Clin Infect Dis. 2021 Nov 2;73(9):e2560-e2568. doi: 10.1093/cid/ciaa754. PMID 32761174
- [Result] George CM, Bhuyian MSI, Thomas ED, Parvin T, Monira S, Zohura F, Hasan MT, Tahmina S, Munmun F, Sack DA, Perin J, Alam M. Psychosocial Factors Mediating the Effect of the CHoBI7 Mobile Health Program on Handwashing With Soap and Household Stored Water Quality: A Randomized Controlled Trial. Health Educ Behav. 2022 Apr;49(2):326-339. doi: 10.1177/1090198120987134. Epub 2021 May 5. PMID 33949243
- [Result] George CM, Zohura F, Teman A, Thomas E, Hasan T, Rana S, Parvin T, Sack DA, Bhuyian SI, Labrique A, Masud J, Winch P, Leontsini E, Zeller K, Begum F, Khan AH, Tahmina S, Munum F, Monira S, Alam M. Formative research for the design of a scalable water, sanitation, and hygiene mobile health program: CHoBI7 mobile health program. BMC Public Health. 2019 Jul 31;19(1):1028. doi: 10.1186/s12889-019-7144-z. PMID 31366398
- [Result] Thomas ED, Zohura F, Hasan MT, Rana MS, Teman A, Parvin T, Masud J, Bhuyian MSI, Hossain MK, Hasan M, Tahmina S, Munmun F, Khan MAH, Monira S, Sack DA, Leontsini E, Winch PJ, Alam M, George CM. Formative research to scale up a handwashing with soap and water treatment intervention for household members of diarrhea patients in health facilities in Dhaka, Bangladesh (CHoBI7 program). BMC Public Health. 2020 Jun 1;20(1):831. doi: 10.1186/s12889-020-08727-0. PMID 32487209
- [Result] Masud J, Islam Bhuyian MS, Kumar Biswas S, Zohura F, Perin J, Papri N, Dil Farzana F, Parvin T, Monira S, Alam M, George CM. Diarrhoeal disease knowledge among diarrhoea patient housholds: findings from the randomised controlled trial of the Cholera-Hospital-Based-Intervention-for-7-days (CHoBI7) mobile health program. Trop Med Int Health. 2020 Aug;25(8):996-1007. doi: 10.1111/tmi.13415. Epub 2020 Jul 21. PMID 32406989
- [Result] Islam Bhuyian MS, Saxton R, Hasan K, Masud J, Zohura F, Monira S, Kumar Biswas S, Tasdik Hasan M, Parvin T, Minhaj I, Md Zillur Rahman K, Papri N, Rashid MU, Sharin L, Teman A, Thomas ED, Alland K, Labrique A, Sack DA, Perin J, Alam M, George CM. Process evaluation for the delivery of a water, sanitation and hygiene mobile health program: findings from the randomised controlled trial of the CHoBI7 mobile health program. Trop Med Int Health. 2020 Aug;25(8):985-995. doi: 10.1111/tmi.13414. Epub 2020 Jul 18. PMID 32406965
- [Result] Zohura F, Bhuyian MSI, Saxton RE, Parvin T, Monira S, Biswas SK, Masud J, Nuzhat S, Papri N, Hasan MT, Thomas ED, Sack D, Perin J, Alam M, George CM. Effect of a water, sanitation and hygiene program on handwashing with soap among household members of diarrhoea patients in healthcare facilities in Bangladesh: a cluster-randomised controlled trial of the CHoBI7 mobile health program. Trop Med Int Health. 2020 Aug;25(8):1008-1015. doi: 10.1111/tmi.13416. Epub 2020 Jul 14. PMID 32406581
- [Result] George CM, Perin J, Parvin T, Bhuyian S, Thomas ED, Monira S, Zohura F, Hasan T, Sack D, Alam M. Effects of a Water, Sanitation and Hygiene Mobile Health Program on Respiratory Illness in Bangladesh: A Cluster-Randomized Controlled Trial of the CHoBI7 Mobile Health Program. Am J Trop Med Hyg. 2022 Jan 10;106(3):979-984. doi: 10.4269/ajtmh.21-0679. PMID 35008045